CLINICAL TRIAL: NCT05556161
Title: Effects of the General Practitioners and Diabetes Specialists Co-management Model for Patients With Type 2 Diabetes in the Community: a Randomized Controlled Trial
Brief Title: Effects of the General Practitioners and Diabetes Specialists Co-management Model for Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: Baoan Central Hospital of Shenzhen (Unknown)
Responsible Party: Principal Investigator, Xiaoxv Yin, PhD, Director of the office of social science and health management, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GPDSCM-T2DM
Record Dates: First submitted 2022-09-22; First posted 2022-09-27 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2023-06

CONDITIONS: Type2diabetes
MeSH Terms: interventions — General Practitioners

STUDY DESIGN:
Intervention Model Description: In parallel arm design, subjects are randomized to one or more study arms and each study arm will be allocated a different intervention. After randomization each subject stays in their assigned treatment arm for the duration of the study. Subjects receive the same treatment throughout the trial. The results are then compared.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant will be blinded of which treatment group subject is assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): The 12-month general practitioners and diabetes specialists co-management will be received by intervention group participants.
  Interventions: Behavioral: General Practitioners and Diabetes Specialists Co-management
- Control group (No Intervention): Routine primary health care will be received by control group participants during the course of the Study.

INTERVENTIONS:
Behavioral: General Practitioners and Diabetes Specialists Co-management — Self-monitoring of blood glucose: Participants will monitor blood glucose with a a free intelligent home blood glucose meter. Then, the intelligent blood glucose meter will upload data to the platform.
  Glycosylated hemoglobin check:
  Cooperative General Practitioner-Specialist Management: Based on the remote monitoring of blood glucose, general practitioners and specialists will jointly carry out management measures including health education, medication adjustment, outpatient consultation, referral, case discussion, etc. for participants.
  Arms: Intervention Group

SUMMARY:
This is a prospective, randomized, parallel, multicenter controlled study to evaluate the effectiveness of the general practitioners and diabetes specialists co-management model for type 2 diabetes. Patients with type 2 diabetes will be randomized to participate in the community general practitioners and diabetes specialists management or serve as controls continuing with routine primary health care. The primary outcome is to observe the HbA1c change.

DETAILED DESCRIPTION:
Aim: This study constructs a general practitioner and diabetes specialist co-management model for patients with type 2 diabetes in the community based on the integration of prevention and treatment strategies. Also, the effectiveness of the model will be evaluated by a parallel randomized controlled trial design to provide theoretical support and empirical evidence for the development of a comprehensive management strategy for patients with type 2 diabetes.

Hypothesis: Compared to the control group, the intervention group receiving co-management by general practitioners and diabetes specialists has a greater improvement in HbA1c, fasting glucose, blood pressure, lipids, BMI, diabetes self-management ability, depression symptoms, diabetes distress, and diabetes complications-related indicators.

Recruiting: This study will recruit patients with type 2 diabetes who have established electronic health records in 5 community healthcare centers affiliated with the Baoan Central Hospital of Shenzhen. General practitioners at the community healthcare centers screen patients with type 2 diabetes under their care who are eligible for the study based on the inclusion and exclusion criteria. Following face-to-face communication, general practitioners explain the study objectives and procedures to patients and obtain their informed consent.

Before the start of the study, unified training will be conducted for the general practitioners involved in the recruitment so that they can clarify the inclusion and exclusion criteria, screening methods, and precautions regarding the study objects.

Randomization Procedure: Members of the research team served as the grouping scheme controllers of the randomization center. The Proc plan procedure of SAS 9.4 statistical software was used to generate random number sequences and grouping schemes according to a 1:1 assignment. For the patients with type 2 diabetes who met the inclusion and exclusion criteria, general practitioners contacted randomization center staff members by telephone according to the patients' order of arrival at the community healthcare center and informed them of the patient's name and ID number. Then the randomization center staff recorded patient information, numbered the patients, and divided them into an intervention group or control group according to the previously generated random number table. Finally, the randomization center staff informed patients' general practitioners of their grouping results.

Study design: The study includes three phases: baseline, intervention, and follow-up. All participants will be divided into an intervention group and a control group after completing the baseline survey. The implementation phase of the intervention will last 18 months. Patients in the intervention group will have daily blood glucose monitoring with a smart home blood glucose meter. Each patient will be assigned a dedicated general practitioner to track the patient's blood glucose monitoring results. Based on the remote monitoring of blood glucose and HbA1c tests, general practitioners and specialists will jointly carry out management measures including health education, medication adjustment, outpatient consultation, referral, and case discussion for participants.

The control group will be routinely treated and followed up by general practitioners according to Chinese clinical guidelines and national norms for basic public health services.

Data collection and management: baseline and follow-up data were collected using questionnaires and physical examination record forms. The collected data was entered into Epidata software and imported into Statistical Analysis System (SAS) 9.4 for analysis. After the end of the experiment, the data will be stored in the database of our research group for a long time.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with type 2 diabetes for over 1 year according to the diagnostic criteria of diabetes formulated by the World Health Organization;
2. Male or female residents aged 18-85 years;
3. HbA1c measured within 6 months before enrollment was 7.0%-10.0%;
4. Lived in the catchment and have established health records for at least 6 months, and have no plans to move out at present;
5. patients used smartphones;
6. Sign the informed consent and participate in the study voluntarily.

Exclusion Criteria:

1. Patients used insulin within 1year before enrollment;
2. patients with type 1 diabetes, Latent autoimmune diabetes of adults(LADA), gestational diabetes, patients with extremely poor islet function (fasting C-peptide < 0.1ng/ml) and patients with special type of diabetes;
3. Patients used continuous glucose monitoring (CGM) in the past 3 months;
4. Patients with serious complications (such as Stage G5 of diabetic nephropathy, severe loss of vision or blindness due to diabetic retinopathy and patients without self-care ability due to diabetic foot amputation).
5. Patients who suffered from serious mental illness or late stage of other serious diseases (such as malignant tumors, acute cardiovascular disease (like stroke, myocardial infarction), serious liver insufficiency, patients with history of diabetic ketoacidosis, patients with alcohol or drug abuse or dependence and patients with a history of cardiac surgery in the last 3 months;
6. Patients with cognitive impairment, or patients unable to use mobile phones to answer calls.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 609 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
HbA1c change | Baseline, 6, and 18 months
  The change of HbA1c during the study. The level of HbA1c in blood measured in %.

SECONDARY OUTCOMES:
Fasting Plasma Glucose | Baseline, 6, and 18 months
  The change of HbA1c during the study.
Total cholesterol | Baseline, 6, and 18 months
  The change of total cholesterol during the study.
Triglycerides | Baseline, 6, and 18 months
  The change of total triglycerides during the study.
LDL-C | Baseline, 6, and 18 months
  The change of LDL-C during the study.
HDL-C | Baseline, 6, and 18 months
  The change of LDL-C during the study.
Blood pressure | Baseline, 6, and 18 months
  The change of blood pressure during the study.
Body Mass Index (BMI) | Baseline, 6, and 18 months
  The change of BMI during the study.
Diabetes self-care activities | Baseline, 6, and 18 months
  Diabetes self-care activities will be measured by the Summary of Diabetes Self-Care Activities (SDSCA) scale. The SDSCA scale measures the frequency of performing diabetes self-care activities, including diet, exercise, blood glucose testing, foot care, and tobacco use over the past 7 days. SDSCA comprises of 11 items and each item's response is rated on 7 point scale ranging from '0' to '7' . A higher score would be the frequency of performing self-care activities.
Diabetes distress | Baseline, 6, and 18 months
  Diabetes distress scores will be measured by the Problem Areas In Diabetes (PAID). The scale ranges from a minimum of 0 (not a problem) to a maximum score of 4 (serious problem). The sum of the five questions provides the participant's score with a score range of minimum score of 0 to a maximum score of 20. A total score of greater than or equal to 8 indicates possible diabetes related emotional distress, with a higher score indicating more significant distress.
Depressive symptoms | Baseline, 6, and 18 months
  Depressive symptoms will be assessed by the Patient Health Questionnaire (PHQ-9). The PHQ-9 is a 9-item scale where respondents indicate how much they are bothered by certain problems on a 4-point scale where 0 = not at all and 3 = nearly every day. Total scores range from 0 to 27 with degree of depression considered minimal for scores between 0-4, mild for scores of 5-9, moderate for scores of 10-14, moderate to severe for scores 15-19, and severe for scores of 20-27.
Self-Efficacy | Baseline, 6, and 18 months
  Participants' self-efficacy level will be measured by the Diabetes Empowerment Scale (DES-SF). The scale consists of 10 items and reports in a 5-points Likert scale. An item checked "strongly agree" receives 5 points; "agree" - 4 points; "neutral" - 3 points; "disagree" - 2 points; and "strongly disagree" receives 1 points. Minimum score is 8, max is 40. Higher scores indicate greater sense of empowerment to self-manage condition.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoxv Yin, Study Director — Huazhong University of Science and Technology
Locations (1):
- Baoan Central Hospital of Shenzhen, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No